CLINICAL TRIAL: NCT05591742
Title: The Effect on Bacterial Composition in Urine, Vagina and Faces After Treatment With Lactobacilli and Its Influence on Recurrent Cystitis in Postmenopausal Women.
Brief Title: Bacterial Composition and Recurrent Cystitis in Postmenopausal Women After Treatment With Lactobacilli.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Caroline S Juhl, Senior registrar, Aalborg University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-20200092
Record Dates: First submitted 2022-10-15; First posted 2022-10-24 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Cystitis Recurrent; Lactobacillus Infection

STUDY DESIGN:
Intervention Model Description: double blinded prospective, randomized cross-over study. Taking place over 6 months with 5 clinical visits.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All (participants, clinical staff, analyzers) are masked until all data have been analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): As it is blinded, no one knows which arm participants enter. After 3 months the other arm is entered.
  Interventions: Other: Placebo Z Cap V-3 Pla
- Femidur (Active Comparator): As it is blinded, no one knows which arm participants enter. After 3 months the other arm is entered.
  Interventions: Dietary Supplement: FEMIDUR®

INTERVENTIONS:
Dietary Supplement: FEMIDUR® — Femidur® consist of 2 vaginal lactobacillis; Lactobacillus rhamnosus GR-1® and Lactobacillus reuteri RC-14®. One tablet a day.
  Placebo Z Cap V-3 Pla; mainly maltodextrin
  Arms: Femidur
Other: Placebo Z Cap V-3 Pla — Consist mainly of maltodextrin. One tablet a day.
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to learn about the effect on the bacterial composition in the microbiome (the body's own bacteria) of urine, vagina and faeces after treatment with lactobacilli (lactobacilli's are a part of the microbiome), and its influence on repeated cystitis in postmenopausal women.

The main questions it aims to answer are:

* Does treatment with lactobacilli change the composition of the urine microbiome in postmenopausal women?
* Does treatment with lactobacilli prevent repeated cystitis in postmenopausal women?

Participants will be followed for 6 months. They will for 3 months receive a look-alike substance that contains no active drug and for the other 3 months tablets with lactobacilli. A computer program will decide what treatment the participant will begin with, and after 3 months she will be receiving the tablets, she did not get first. This way all participants receive both type of tablets and can be their own control. What type of tablet the participants is taking is unknown to both clinical staff and participants.

The participants will come to the hospital for start-up, and every 1,5 moths for the next 6 months.

They deliver

* faeces sample
* urine tests
* vaginal swab

each time they are seen.

When entering the study, they also complete health care questions on medication, earlier surgery, alcohol, tobacco, childbirths, weight, height etc. They make a drinking and voiding diary 3 times over the 6 months.

When the study is over, alle the samples of faeces, urine and the vaginal swab will undergo analyzation for the bacterial composition in the microbiome, and differences in the microbiome when taking lactobacilli or not will be examined. The urine sample is controlled for bacteria known to give cystitis, and the influence on repeated cystitis will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women
* if hysterectomy before menopause, then age of >60 years
* verified diagnose of recurrent cystitis. (two in 6 months or 3 in a year, verified by cultivation)
* able to speak and write Danish

Exclusion Criteria:

* vaginal prolapse with symptoms
* residual urine over 150 ml
* bladder diseases
* profylactic antibiotics
* probiotics
* bladder cancer
* genital cancer.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — it can only be females with chromosome XX due to influence on hormones' and the length of urinary tract.
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
The change in the urine microbiome among postmenopausal women when treated with lactobacillis | after study completion, an average of 1.5 year
  The micobiom will be analysed by 16s rRNA sequencing.
The change in the urine microbiome among postmenopausal women when treated with lactobacillis | after study completion, an average of 1.5 year
  Operational taxonomic unit (OTU) richness
The change in the urine microbiome among postmenopausal women when treated with lactobacillis | after study completion, an average of 1.5 year
  Shannon Index, as expression for the alpha diversity
The change in the urine microbiome among postmenopausal women when treated with lactobacillis | after study completion, an average of 1.5 year
  Beta diversity by means of PCA plots

SECONDARY OUTCOMES:
episodes of UTI | after study completion, an average of 2 months
  in numbers over time.
changes in vaginal micobiome | after study completion, an average of 1.5 year
  The micobiom will be analysed by 16s rRNA sequencing.
changes in vaginal micobiome | after study completion, an average of 1.5 year
  Operational taxonomic unit (OTU) richness
changes in vaginal micobiome | after study completion, an average of 1.5 year
  Shannon Index, as expression for the alpha diversity
changes in vaginal micobiome | after study completion, an average of 1.5 year
  Beta diversity by means of PCA plots
Changes in fecal microbiome | after study completion, an average of 1.5 year
  The micobiom will be analysed by 16s rRNA sequencing.
Changes in fecal microbiome | after study completion, an average of 1.5 year
  Operational taxonomic unit (OTU) richness
Changes in fecal microbiome | after study completion, an average of 1.5 year
  Shannon Index, as expression for the alpha diversity
Changes in fecal microbiome | after study completion, an average of 1.5 year
  Beta diversity by means of PCA plots

CONTACTS AND LOCATIONS:
Overall Officials: Caroline S Juhl, Principal Investigator — Aalborg University Hospital
Locations (1):
- AalborgH, Aalborg, Region Nord, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT05591742/Prot_SAP_000.pdf